CLINICAL TRIAL: NCT05927454
Title: Cohorte d'Adultes et d'Enfants Avec Maladie de Still
Brief Title: Acostill ( RaDiCo Cohort) (RaDiCo Acostill)
Acronym: Acostill
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-48
Record Dates: First submitted 2021-12-20; First posted 2023-07-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Still Disease; Still's Disease, Adult-Onset; Still Disease, Juvenile Onset
Keywords: Still Disease; Rare disease; Diagnostic markers; Prognostic markers; New therapies
MeSH Terms: conditions — Arthritis, Juvenile; Still's Disease, Adult-Onset; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adult Onset Still Disease (AOSD) and Systemic onset Juvenile Idiopathic Arthritis (SoJIA) are two rare multifactorial diseases associated with systemic inflammation. These two forms AOSD and SoJIA are considered to be two facets of the same syndrome, combining four cardinal symptoms [hectic fever> 39 °, arthralgia or arthritis, skin rash, a leukocyte formula with more than 80% of neutrophils]; lymphadenopathy and splenomegaly may also be found. There is an important biological inflammatory syndrome with elevation of the reactive C protein, of serum ferritin with a dramatic drop in the glycosylated fraction. The incidence of the disease is low, around 0.1/100,000 for adults and 0.6/100,000 for children. Its prevalence is approximately 1 to 3/100,000 and 3/100,000 for children, so there are approximately 500 to 1,500 adults and 450 children affected in France. It is subdivided into pediatric and adult forms according to the age of onset before or after 16 years. The prognosis of the disease is functional and vital. Macrophage activation syndrome (SAM) is frequently associated with either the onset of the disease or the initiation of treatment or concomitantly with viral reactivation. The course over time has mainly been studied in children and is variable: regression, course by flare-ups with term regression and chronic joint development. In adults we can also observe these 3 evolutionary modes. However, differences seem to exist between AOSD and SoJIA.

The various clinical questions posed by this disease are as follows:

* Why does it differentially affect two age groups of the population?
* Why is the clinical expression heterogeneous with pure systemic or articular forms, the frequency of SAM, and rare organ damage?
* Why is the evolution over time different with resolving monocyclic forms or polycyclic forms and sometimes chronic evolutions?

These differences could be explained by distinct underlying pathogenic mechanisms. But at present, the pathophysiology of this entity remains unknown, although several hypotheses can be formulated involving several pathophysiological pathways.

The pathogenesis of Still's disease has not yet been elucidated but there is a significant inflammatory reaction without the production of autoantibodies, which makes this disease a form of autoinflammatory syndrome with abnormalities of the innate immunity (activation of macrophages, strong elevations of pro-inflammatory cytokines: interleukins 1 and 18, possible abnormalities of inflammasomes and NK cells). The treatment is based on anti-inflammatory drugs, corticosteroids with the usefulness of methotrexate and anti-TNF in the event of significant joint damage. Interleukin 1 and 6 inhibitors have been shown to be effective in this disease. In adults and children, there are forms that are refractory to treatment, with a risk of AA amyloidosis for these patients.

The expected outcomes of this work are to improve knowledge of Still disease and patient management on the following aspects:

* Comparison of pediatric and adult forms (which has never been done on a large number of patients),
* Better understanding of the pathogenic mechanisms of the disease,
* The identification of early diagnostic/prognostic markers,
* The possibility of promoting the evaluation of new therapies to come thanks to the constitution of an active file of patients with a standardized follow-up.

The ACOSTILL study group is thus a unique collaboration of adult clinicians (rheumatologists and internists) and pediatricians, who have decided to unite their efforts to increase knowledge about the pathogenesis of Still disease in order to better understand the disease and improve care pathways. Many of them participated in the development of the national diagnostic and care protocol published in 2018.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 16 (age> 16) meeting the diagnostic criteria of Yamaguchi or Fautrel criteria (appendix 5)
* Aged 16 years or less (age ≤16 years) fulfilling the 2001 criteria for ILAR systemic form of juvenile idiopathic arthritis
* Having signed a consent to participate in the cohort and in the collection of clinical and biological data; in accordance with the regulations, for patients who are minors or adults who are protected, the non-opposition of the legal representatives will be sought.
* Affiliated to the "Régime National d'Assurance Maladie".

Exclusion Criteria:

* Other cause of relapsing infectious fever (such as tuberculosis, toxoplasmosis, deep abscesses, viroses, sepsis) or tumor (such as lymphomas)
* Other defined inflammatory rheumatism such as rheumatoid arthritis, psoriatic arthritis, spondyloarthropathies.
* Autoimmune inflammatory disease (systemic lupus erythematosus), granulomatosis (sarcoidosis, Blau syndrome), vasculitis (Behçet's disease, nodular arteritis), polymyositis and dermatomyositis.
* Well-defined auto-inflammatory syndromes with unambiguous mutations, such as familial Mediterranean fever, cryopyrinopathies, TRAPS, mevalonate kinase deficiency.
* Known macrophage activation syndromes of genetic origin.
* Patients unable to understand the information leaflet and sign the informed consent form
* Patients not affiliated to the "Régime National d'Assurance Maladie"

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In order to reflect the reality of daily practice, all pediatric and adult patients already diagnosed and monitored (prevalent patients) or newly diagnosed (incident patients) in one of the French Rare Disease Reference Center or Rare Disease Competence Center will be invited. to participate in the study. In order to document the improvement in patient care, morbidity and mortality through the implementation of the PNDS Still, deceased patients may be included in the cohort.
  The objective is to recruit a minimum of 200 adult patients and 300 pediatric patients so that the study has sufficient statistical power. The stratification of patients is made into 4 subgroups according to the form of the pathology:
  * Pediatric (juvenile arthritis systemic idiopathic)
  * Adult monocyclic (approximately 30% of cases)
  * Adult intermittent or polycyclic (30%)
  * Adult persistent or chronic (40%)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
General signs of the disease | Through study completion, at 1 year, 2 year, 3 year, 4 year, 5 year
Clinical signs of the disease | Through study completion, at 1 year, 2 year, 3 year, 4 year, 5 year
Biological results | Through study completion, at 1 year, 2 year, 3 year, 4 year, 5 year
- The impact of the disease on the patient's daily life | Through study completion, at 1 year, 2 year, 3 year, 4 year, 5 year

SECONDARY OUTCOMES:
Quality of life scores | Through study completion, at 1 year, 2 year, 3 year, 4 year, 5 year
  Measurement of changes in quality of life scores obtained throughout the study
AIDAI scores | Through study completion, at 1 year, 2 year, 3 year, 4 year, 5 year
  Measurement of the individual evolution of the AIDAI (Validation of the Auto-Inflammatory Diseases Activity Index) scores obtained throughout the study
Prospective biomarkers | Through study completion, at 1 year, 2 year, 3 year, 4 year, 5 year
  Search for an association between the prospective biomarkers (pro and anti-inflammatory cytokines, AAS, S100 protein, soluble CD163, ferritinemia and glycosylated ferritinemia) and the diagnosis made (different clinical forms of Still's disease)
Presence of autoinflammatory disease in relatives | Through study completion, at 1 year, 2 year, 3 year, 4 year, 5 year
  Construction of a family tree based on the presence of autoinflammatory disease in relatives

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Georgin-Lavialle, PHD, Principal Investigator — INSERM U933
Locations (1):
- RaDiCo-AcoStill, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided